CLINICAL TRIAL: NCT05055739
Title: Comparative Study Between Sternal Closure With Sternalock® Blue Versus Steel Wire Submitted To Bilateral Anterior Transsternal Thoracotomy (Clamshell) For Bilateral Lung Transplant
Acronym: LungTx-Lock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Paulo Manuel Pêgo Fernandes, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University of Sao Paulo
Record Dates: First submitted 2021-05-26; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Lung; Lung Transplant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SW (Experimental): Patients undergoing sternal closure with steel wires
  Interventions: Device: Rigid plate X steel wires
- RP (Experimental): Patients undergoing sternal closure with a rigid plate
  Interventions: Device: Rigid plate X steel wires

INTERVENTIONS:
Device: Rigid plate X steel wires — Compare the sternal alignment between the fixation with rigid plate X steel wires.

SUMMARY:
This will be a prospective, randomized clinical trial, comparing the sternal alignment between the fixation with rigid plate X steel wires. Patients over 18 years of age, belonging to the lung transplant line in the State of São Paulo, who will undergo bilateral lung transplantation will be studied.

ELIGIBILITY:
Inclusion Criteria:

1. Above 18 years of age;
2. Belonging to the transplant queue of InCor;
3. Eligible for sequential bilateral lung transplantation submitted to clamshell incision;

Exclusion Criteria:

1. Patients undergoing a new surgical procedure after lung transplantation with the need to manipulate the steel wires or the sternal fixation plate other than for osteomyelitis;
2. Intraoperative death;
3. Patients who have undergone unilateral lung transplantation or have not undergone a clamshell incision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Sternal Alignment | 1 month
  Sternal alignment will be analyzed through cross-sections of chest computed tomography by a certified radiologist.
  Two parameters will be used for sternal alignment:
  Misalignment:
  1. Significant:> 3mm;
  2. Non-significant: ≤3mm
  Deviation:
  1. Grade 1: ≤50%
  2. Grade 2:> 50%
Sternal Alignment | 3 months
  Sternal alignment will be analyzed through cross-sections of chest computed tomography by a certified radiologist.
  Two parameters will be used for sternal alignment:
  Misalignment:
  1. Significant:> 3mm;
  2. Non-significant: ≤3mm
  Deviation:
  1. Grade 1: ≤50%
  2. Grade 2:> 50%
Sternal Alignment | 6 months
  Sternal alignment will be analyzed through cross-sections of chest computed tomography by a certified radiologist.
  Two parameters will be used for sternal alignment:
  Misalignment:
  1. Significant:> 3mm;
  2. Non-significant: ≤3mm
  Deviation:
  1. Grade 1: ≤50%
  2. Grade 2:> 50%

SECONDARY OUTCOMES:
Bone healing | 1 month
  Bone healing will be analyzed through cross-sections of chest computed tomography by a certified radiologist.
  • The degree of bone healing will be classified into 6 levels: 0- (A) No signs of consolidation (no clear consolidation, no union, sternal separation)
  1. (B) Minimal consolidation (sternal separation, lack of bone bridge)
  2. (C) Median consolidation (sternal separation with some trace of bone bridge, immature bone formation)
  3. (D) Moderate consolidation (partial bone connection indicating sternal stability)
  4. (E) Partial synthesis (significant bone bridge)
  5. (F) Complete synthesis (complete bone bridge)
Bone healing | 3 months
  Bone healing will be analyzed through cross-sections of chest computed tomography by a certified radiologist.
  • The degree of bone healing will be classified into 6 levels: 0- (A) No signs of consolidation (no clear consolidation, no union, sternal separation)
  1. (B) Minimal consolidation (sternal separation, lack of bone bridge)
  2. (C) Median consolidation (sternal separation with some trace of bone bridge, immature bone formation)
  3. (D) Moderate consolidation (partial bone connection indicating sternal stability)
  4. (E) Partial synthesis (significant bone bridge)
  5. (F) Complete synthesis (complete bone bridge)
Bone healing | 6 months
  Bone healing will be analyzed through cross-sections of chest computed tomography by a certified radiologist.
  • The degree of bone healing will be classified into 6 levels: 0- (A) No signs of consolidation (no clear consolidation, no union, sternal separation)
  1. (B) Minimal consolidation (sternal separation, lack of bone bridge)
  2. (C) Median consolidation (sternal separation with some trace of bone bridge, immature bone formation)
  3. (D) Moderate consolidation (partial bone connection indicating sternal stability)
  4. (E) Partial synthesis (significant bone bridge)
  5. (F) Complete synthesis (complete bone bridge)
Pain | 1 month
  The patients' postoperative pain will be assessed according to the Pain Score (Pain Score).
Pain | 3 months
  The patients' postoperative pain will be assessed according to the Pain Score (Pain Score).
Pain | 6 months
  The patients' postoperative pain will be assessed according to the Pain Score (Pain Score).
Time to close the Rib cage | 1 month
  Time to close the Rib cage will be measured from the insertion of the last chest drain until the total closure of the skin of the thorax.
Time to close the Rib cage | 3 months
  Time to close the Rib cage will be measured from the insertion of the last chest drain until the total closure of the skin of the thorax.
Time to close the Rib cage | 6 months
  Time to close the Rib cage will be measured from the insertion of the last chest drain until the total closure of the skin of the thorax.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coração - HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No